CLINICAL TRIAL: NCT00623363
Title: A Double-Blind, Placebo-Controlled, Preliminary Study of the Efficacy, Safety, and Tolerability of Intravenous SUN N4057 in Patients With Motor Complications Associated With Parkinson's Disease
Brief Title: Preliminary Study of Piclozotan in Patients With Motor Complications Associated With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASBI-501
Record Dates: First submitted 2008-01-02; First posted 2008-02-26 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; motor complications; dyskinesia; Motor complications associated with Parkinson's
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — Piclozotan; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- piclozotan (Active Comparator): Participants will be randomized to receive two 12-hour intravenous (IV) infusions of piclozotan administered at a plasma level of 30 ng/mL over 2 inpatient days.
  Interventions: Drug: piclozotan
- 0.9 % sodium chloride (normal saline) (Placebo Comparator): Participants will be randomized to receive two 12-hour intravenous (IV) infusions of 0.9 % sodium chloride (normal saline) administered at a plasma level of 30 ng/mL over 2 inpatient days.
  Interventions: Drug: 0.9% sodium chloride (normal saline)

INTERVENTIONS:
Drug: piclozotan — piclozotan, intravenous (IV) infusion
  Other Names: SUN N4057
  Arms: piclozotan
Drug: 0.9% sodium chloride (normal saline) — 0.9% sodium chloride (normal saline) intravenous (IV) infusion
  Arms: 0.9 % sodium chloride (normal saline)

SUMMARY:
The purpose of this study is to obtain preliminary information on the effect of piclozotan on motor complications associated with Parkinson's Disease.

ELIGIBILITY:
Main Inclusion Criteria:

* Idiopathic Parkinson's disease for at least 5 years
* Presence of motor fluctuations and dyskinesia
* Stable regimen of levodopa/carbidopa for 30 days
* At least 25% response/improvement in Unified Parkinson's Disease Rating Scale (UPDRS) part III scores after dosing with regular Parkinson's disease (PD) medications
* Mini-Mental State Examination (MMSE) score of 25 or higher

Main Exclusion Criteria:

* Atypical or secondary parkinsonism.
* Prior use of neuroleptic agents.
* History of intracranial procedures for PD.
* Active psychosis.
* History of drug or alcohol abuse in past 12 months.
* Cardiac conduction system abnormality.
* Predisposing medical condition that causes nausea or vomiting or routine use of an anti-emetic.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-07-13 (Actual); Primary Completion 2008-07-17 (Actual); Study Completion 2008-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (7):
- United States (5):
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - University of South Florida, Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Emory University--Wesley Woods Health Center, Atlanta, Georgia
  - UMDNJ-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Suny Downstate Medical Center, Brooklyn, New York
- Hospital Multimedica, Guatemala City, Guatemala
- Hospital Clinic of Neurology and Psychiatry Oradea, Oradea, Romania

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 27 participants who met all inclusion criteria and no exclusion criteria were enrolled in the study at 4 clinic sites in the United States of America (USA), 1 in Guatemala, and 1 in Romania.
Groups:
- Placebo: Participants with Parkinson's disease who were administered two 12-hour IV infusions of 0.9% sodium chloride (normal saline) placebo over 2 inpatient days.
- SUN N4057: Participants with Parkinson's disease who were administered two 12-hour IV infusions of SUN N4057 (piclozotan) over 2 inpatient days.
Period: Overall Study
Arm/Group | Placebo | SUN N4057
Started | 7 | 20
Completed | 5 | 18
Not Completed | 2 | 2
Not completed — Adverse Event | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed using the Safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SUN N4057 | Total
Number analyzed (Participants) | 7 | 18 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (9.47) | 59.3 (11.51) | 59.9 (10.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 5 | 14 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 13 | 17
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 6 | 9
  More than one race | NA — More than one race was not assessed. | NA — More than one race was not assessed. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported | 3 | 12 | 15
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9
  Guatemala | 3 | 13 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Percentage of "On" Time Without Dyskinesia Averaged Over Days 1 and 2 in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: Improvement in motor complications associated with Parkinson's disease are measured as "on" (good medication response); OR "on with dyskinesia" (good medication response, but with superimposed involuntary movements that interfere with activities), OR "off" (poor medication response).
Time Frame: Baseline (Day-7) up to 2 days post-dose.
Population: The percentage of "on" time without dyskinesia was assessed using the modified intent-to-treat (MITT) population.
Measure: Mean (Standard Deviation); unit: percentage of on time
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
percentage of on time
  Baseline (Day -7) | 12.50 (10.21) | 18.75 (22.38)
  Average of Days 1 and 2 | 17.86 (25.37) | 36.11 (26.99)
  Change from Baseline | 5.36 (20.23) | 17.36 (24.96)
Statistical Analysis 1: Comparison: SUN N4057; Baseline (Day -7); Test type: Superiority; p = 0.503, Monte Carlo estimates
Statistical Analysis 2: Comparison: Placebo; Average of Days 1 and 2; Test type: Superiority; Least Squares (LS) Mean = 20.60, 95% CI 2-sided [1.82 to 39.37]
Statistical Analysis 3: Comparison: Placebo; Change from Baseline; Test type: Superiority; Least Squares (LS) Mean = 3.60, 95% CI 2-sided [-15.18 to 22.37]
Statistical Analysis 4: Comparison: SUN N4057; Average of Days 1 and 2; Test type: Superiority; Least Squares (LS) Mean = 36.59, 95% CI 2-sided [24.04 to 49.14]
Statistical Analysis 5: Comparison: SUN N4057; Change from Baseline; Test type: Superiority; p = 0.160, ANCOVA; Least Squares (LS) Mean = 19.59, 95% CI 2-sided [7.04 to 32.14]

2. Secondary Outcome: Change From Baseline up to Day 2 in the Percentage of "on" Time Without Dyskinesia, as Assessed Over Hours 1 to 8 for Each Time Point in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: as for outcome 1
Time Frame: Baseline (Day -7), Day 1, and Day 2 post-dose.
Population: The percentage of "on" time without dyskinesia was assessed using the modified intent-to-treat (MITT) population.
Measure: Mean (Standard Deviation); unit: percentage of on time
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
percentage of on time
  Baseline (Day -7) | 12.50 (10.21) | 18.75 (22.38)
  Day 1 | 23.21 (33.41) | 31.25 (30.39)
  Change from Baseline to Day 1 | 10.71 (29.25) | 12.50 (25.73)
  Day 2 | 12.50 (19.09) | 40.97 (35.04)
  Change from Baseline to Day 2 | 0.00 (12.50) | 22.22 (35.76)

3. Secondary Outcome: Percentage of "on" Time With Dyskinesia at Baseline up to Day 2, and the Change From Baseline in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: Improvement in motor complications associated with Parkinson's disease are measured as "on" (good medication response); OR "on with dyskinesia" (good medication response, but with superimposed involuntary movements that interfere with activities), OR "off" (poor medication response). Negative values indicate a decrease in "on" time from baseline to measured time point.
Time Frame: Baseline (Day -7), Day 1, and Day 2 post-dose.
Population: The percentage of "on" time with dyskinesia was assessed using the modified intent-to-treat (MITT) population.
Measure: Mean (Standard Deviation); unit: percentage of on time
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
percentage of on time
  Baseline (Day -7) | 78.57 (13.91) | 60.42 (26.17)
  Day 1 | 55.36 (41.37) | 48.61 (27.75)
  Change from Baseline to Day 1 | -23.21 (32.62) | -11.81 (31.64)
  Day 2 | 64.29 (28.35) | 49.31 (33.89)
  Change from Baseline to Day 2 | -14.29 (19.67) | -11.11 (32.90)

4. Secondary Outcome: Percentage of "on" Time With Dyskinesia for the Average of Days 1 and 2, and the Change From Baseline in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: as for outcome 3
Time Frame: Baseline (Day -7), Day 1, and Day 2 post-dose.
Population: The percentage of "on" time with dyskinesia was assessed using the modified intent-to-treat (MITT) population.
Measure: Mean (Standard Deviation); unit: percentage of on time
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
percentage of on time
  Average of Days 1 and 2 | 59.82 (34.40) | 48.96 (22.51)
  Change from Baseline | -18.75 (25.52) | -11.46 (24.28)

5. Secondary Outcome: Percentage of "on" Time With or Without Dyskinesia at Baseline up to Day 2, and the Change From Baseline in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: as for outcome 3
Time Frame: Baseline (Day -7), Day 1 and Day 2 post-dose.
Population: The percentage of "on" time with or without dyskinesia was assessed using the modified intent-to-treat (MITT) population.
Measure: Mean (Standard Deviation); unit: percentage of on time
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
percentage of on time
  Baseline (Day -7) | 91.07 (15.67) | 79.17 (19.65)
  Day 1 | 78.57 (26.73) | 79.86 (25.05)
  Change from Baseline to Day 1 | -12.50 (19.09) | 0.69 (24.81)
  Day 2 | 76.79 (29.25) | 90.28 (18.47)
  Change from Baseline to Day 2 | -14.29 (20.95) | 11.11 (20.06)

6. Secondary Outcome: Percentage of "on" Time With or Without Dyskinesia for the Average of Days 1 and 2, and the Change From Baseline in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: as for outcome 3
Time Frame: Baseline (Day -7), Day 1 and Day 2 post-dose.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percentage of on time
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
percentage of on time
  Average of Days 1 and 2 | 77.68 (27.92) | 85.07 (20.47)
  Change from Baseline | -13.39 (19.91) | 5.90 (21.06)

7. Secondary Outcome: Percentage of "Off" Time at Baseline up to Day 2, and the Change From Baseline in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: Improvement in motor complications associated with Parkinson's disease are measured as "on" (good medication response); OR "on with dyskinesia" (good medication response, but with superimposed involuntary movements that interfere with activities), OR "off" (poor medication response). Negative values indicate a decrease in "off" time from baseline to measured time point.
Time Frame: Baseline (Day -7), Day 1, and Day 2 post-dose.
Population: The percentage of "off" time was assessed using the modified intent-to-treat (MITT) population.
Measure: Mean (Standard Deviation); unit: percentage of off time
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
percentage of off time
  Baseline (Day -7) | 8.93 (15.67) | 20.83 (19.65)
  Day 1 | 21.43 (26.73) | 20.14 (25.05)
  Change from Baseline to Day 1 | 12.50 (10.09) | -0.69 (24.81)
  Day 2 | 23.21 (29.25) | 9.72 (18.47)
  Change from Baseline to Day 2 | 14.29 (20.95) | -11.11 (20.06)

8. Secondary Outcome: Percentage of "Off" Time for the Average of Days 1 and 2, and the Change From Baseline in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: as for outcome 7
Time Frame: Baseline (Day -7), Day 1, and Day 2 post-dose.
Population: The percentage of "off" time was assessed using the modified intent-to-treat (MITT) population.
Measure: Mean (Standard Deviation); unit: percentage of off time
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
percentage of off time
  Average of Days 1 and 2 | 22.32 (27.92) | 14.93 (20.47)
  Change from Baseline | 13.39 (19.91) | -5.90 (21.06)

9. Secondary Outcome: Change From Baseline up to Day 2 in the Average Abnormal Involuntary Movement Scale (AIMS) Total Score in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: The Abnormal Involuntary Movement Scale (AIMS) is an assessment of dyskinesia in patients with movement disorders. The AIMS was originally developed to assess neuroleptic-induced extrapyramidal symptoms but has also been applied to the assessment of dyskinesia in patients with Parkinson's disease. AIMS questions 1 to 7 rate the degree of dyskinesia on a 0 to 4 scale in the extremities, trunk, and face, where 0 is no dyskinesia (better outcome) and 4 is severe dyskinesia (worse outcome). The total score range is 0 (better outcome) to 28 (worse outcome). Higher scores indicate a worse outcome.
Time Frame: Baseline (Day -7), Day 1, and Day 2 post-dose.
Population: The average abnormal involuntary movement scale was assessed using the modified intent-to-treat (MITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
units on a scale
  Baseline (Day -7) | 5.80 (1.94) | 4.31 (2.28)
  Day 1 | 3.11 (3.74) | 2.60 (2.04)
  Change from Baseline to Day 1 | -2.70 (3.16) | -1.70 (3.16)
  Day 2 | 2.98 (2.43) | 2.66 (1.91)
  Change from Baseline to Day 2 | -2.82 (2.82) | -1.65 (2.31)

10. Secondary Outcome: Average of Days 1 and 2 in the Average Abnormal Involuntary Movement Scale (AIMS) Total Score in Participants Treated With SUN N4057 and Those Treated With a Placebo
Description: as for outcome 9
Time Frame: Day 1 and Day 2 post-dose.
Population: The average abnormal involuntary movement scale was assessed using the modified intent-to-treat (MITT) population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
units on a scale
  Average of Days 1 and 2 | 3.04 (3.00) | 2.63 (1.49)
  Change from Baseline | -2.76 (2.83) | -1.67 (2.44)

11. Secondary Outcome: Mean SUN N4057 Plasma Concentrations Over Time Following Treatment With SUN N4057
Description: The mean concentration of study drug, SUN N4057, in participant blood plasma samples drawn during infusions.
Time Frame: Day 1 pre-dose (Hour 0), 1 hour, 6 hours, 12 hours; Day 2 pre-dose (Hour 24), 1 hour (Hour 25), 6 hours (Hour 30), 12 hours (Hour 36), and Day 3 Hour 0 (Hour 48) post-dose.
Population: Mean plasma concentrations were assessed using the pharmacokinetic (PK) population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SUN N4057
Number analyzed (Participants) | 17
ng/mL
  Day 1: Hour 0 | 0.00 (0.00)
  Day Day 1: Hour 1: number analyzed (Participants) | 16
  Day Day 1: Hour 1 | 33.40 (9.71)
  Day 1: Hour 6 | 28.34 (9.19)
  Day 1: Hour 12 | 32.46 (12.26)
  Day 2: Hour 0 | 11.26 (4.66)
  Day 2: Hour 1 | 31.91 (9.52)
  Day 2: Hour 6 | 26.85 (7.92)
  Day 2: Hour 12 | 37.75 (33.02)
  Day 3: Hour 0 | 12.65 (6.08)

12. Secondary Outcome: Mean SUN N4057 Plasma Pharmacokinetic Parameter of Observed Maximum Concentration (Cmax) Following Treatment With SUN N4057
Description: Cmax is the observed maximum concentration of SUN N4057 in the participant blood plasma sample after drug administration.
Time Frame: Baseline (Day 1 pre-dose) up to Hour 24, and Hour 48 post-dose.
Population: Cmax was assessed using the pharmacokinetic (PK) population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SUN N4057
Number analyzed (Participants) | 17
ng/mL | 46.95 (31.46)

13. Secondary Outcome: Mean SUN N4057 Plasma Pharmacokinetic Parameter of Observed Minimum Concentration (Cmin) Following Treatment With SUN N4057
Description: Cmin is the observed minimum concentration of SUN N4057 in the participant blood plasma sample after drug administration. Average of C24 and C48 [ie, 24 hours after the initiation of infusion on Days 1 and 2. Cmin = average of (C24 and C48)
Time Frame: Day 1 pre-dose (Hour 0) up to Hour 24, and Hour 48 post-dose.
Population: Cmin was assessed using the pharmacokinetic (PK) population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SUN N4057
Number analyzed (Participants) | 17
ng/mL | 11.95 (5.30)

14. Secondary Outcome: Mean SUN N4057 Plasma Pharmacokinetic Parameter of Observed Mean Concentration (Caverage) Following Treatment With SUN N4057
Description: Caverage is the mean concentration of SUN N4057 in the participant blood plasma sample obtained from the observed concentrations during the 2-day drug infusions (average of C1, C6, C12, C25, C30, and C36 [ie, Hours 1, 6, 12, 25, 30, and 36 after the initiation of infusion on Day 1]). Caverage = average of (C1, C6, C12, C25, C30, and C36)
Time Frame: Day 1 at 1 hour, 6 hours, and12 hours; Day 2 at 25 hours, 30 hours, and 36 hours post-dose.
Population: Caverage was assessed using the pharmacokinetic (PK) population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SUN N4057
Number analyzed (Participants) | 17
ng/mL | 31.91 (8.96)

15. Secondary Outcome: Mean SUN N4057 Pharmacokinetic Parameter of Area Under the Drug Concentration vs Time Curve (AUCt) Following Treatment With SUN N4057
Description: AUCt is defined as the area under the drug concentration vs time curve from zero up to the last sampling point with a quantifiable drug concentration which is above the lower limit of quantification.
Time Frame: Baseline (Day 1 pre-dose) up to Hour 0, Hour 1, Hour 6, Hour 12, Hour 24, Hour 25, Hour 30, Hour 36, and Hour 48 post-dose.
Population: AUCt was assessed using the pharmacokinetic (PK) population.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SUN N4057
Number analyzed (Participants) | 17
ng*hr/mL | 1271.20 (409.39)

16. Secondary Outcome: Treatment-Related Treatment-Emergent Adverse Events Reported Following Treatment With SUN N4057 or Placebo
Description: A treatment-emergent adverse event (TEAE) was defined as an Adverse Event (AE) that was new in onset or aggravated in severity or frequency following administration of the investigational agent. This included any change from the screening physical examination findings or results of diagnostic procedures (eg, laboratory test, ECG) that were clinically significant, eg, required diagnostic or therapeutic intervention beyond confirmation alone.
Time Frame: Baseline up to Day 16 post-dose, up to approximately a total 12 months.
Population: Treatment-emergent adverse events (TEAEs) were assessed using the Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SUN N4057
Number analyzed (Participants) | 7 | 18
Participants
  Patients with Any TEAE | 6 | 17
  Nausea | 2 | 12
  Dizziness | 0 | 8
  Hypertension | 0 | 7
  Vomiting | 0 | 7
  Disorientation | 1 | 3
  Headache | 0 | 4
  Dyskinesia | 1 | 2
  Hyperhidrosis | 0 | 3
  Blood Pressure increased | 2 | 0
  Cold sweat | 0 | 2
  Abdominal pain | 0 | 1
  Arrhythmia | 1 | 0
  Asthenia | 0 | 1
  Bundle branch block right | 1 | 0
  Chills | 0 | 1
  Confusional state | 0 | 1
  Dizziness postural | 0 | 1
  Ear pain | 0 | 1
  Electrocardiogram abnormal | 0 | 1
  Electrocardiogram QT prolonged | 1 | 0
  Fecal incontinence | 0 | 1
  Flushing | 0 | 1
  Heart rate increased | 1 | 0
  Hypotension | 0 | 1
  Muscle spasms | 1 | 0
  Nightmare | 0 | 1
  Paresthesia | 0 | 1
  Peripheral coldness | 0 | 1
  Somnolence | 0 | 1
  Tachycardia | 0 | 1
  Tremor | 0 | 1
  Vision blurred | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were assessed from the date the informed consent was given to Day 16 post-dose, up to approximately a total of 12 months.
Description: A treatment-emergent adverse event (TEAE) was defined as an Adverse Event (AE) that was new in onset or aggravated in severity or frequency following administration of the investigational agent. This included any change from the screening physical examination findings or results of diagnostic procedures (eg, laboratory test, ECG) that were clinically significant, eg, required diagnostic or therapeutic intervention beyond confirmation alone.
Arm/Group | Placebo | SUN N4057
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/18
Other Adverse Events (participants affected / at risk) | 6/7 | 17/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | SUN N4057 (N=18)
Nausea (Gastrointestinal disorders) | 2 | 12
Dizziness (Nervous system disorders) | 0 | 8
Hypertension (Vascular disorders) | 0 | 7
Vomiting (Gastrointestinal disorders) | 0 | 7
Disorientation (Psychiatric disorders) | 1 | 4
Headache (Nervous system disorders) | 0 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 4
Dyskinesia (Nervous system disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Blood pressure increased (Investigations) | 2 | 0
Cold sweat (General disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0
Chills (Musculoskeletal and connective tissue disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Electrocardiogram abnormal (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Fecal incontinence (Gastrointestinal disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Injection site extravasation (Injury, poisoning and procedural complications) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No